CLINICAL TRIAL: NCT00466063
Title: A 5 Year Observational Study (Registry) of Children Aged 2 to <6 Years at Enrollment With Transfusional Hemosiderosis Treated With Deferasirox
Brief Title: ENTRUST, a 5 Year Surveillance of Children Aged 2 to <6 Years With Transfusional Iron Overload Treated With Deferasirox
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CICL670A2411
Record Dates: First submitted 2007-04-25; First posted 2007-04-27 (Estimated); Last update posted 2015-12-29 (Estimated); Status verified 2015-12

CONDITIONS: Anemia
Keywords: Iron overload; children; deferasirox; Transfusion-dependent anemia
MeSH Terms: conditions — Anemia; Iron Overload | interventions — Deferasirox

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- ICL670: ICL670
  Interventions: Drug: Deferasirox

INTERVENTIONS:
Drug: Deferasirox

SUMMARY:
This registry will evaluate long-term safety and efficacy of deferasirox in children with transfusional iron overload.

ELIGIBILITY:
Inclusion Criteria:

* History of transfusion-dependent anemia.
* History of iron overload

Exclusion Criteria:

* Patients with non-transfusional hemosiderosis.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 200 unselected children aged from 2 to <6 years at enrolment with chronic iron overload due to repeated blood transfusions. The participating countries were selected on the basis of both a high incidence of young children with thalassemia or other transfusion dependent anemias and on the basis that the drug is approved and 'on the market' in the country selected.
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2007-05; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Safety - renal and hepatic function monitoring. | 5 years

SECONDARY OUTCOMES:
Adverse events | 5 years
Longitudinal ferritin levels | 5 years
Assessment of auditory and ophthalmologic status | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (23):
- United States (23):
  - University of South Alabama Medical Center, Mobile, Alabama
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Stanford University Medical Center, Stanford, California
  - MD Anderson Cancer Center - Orlando, Orlando, Florida
  - St. Joseph's Children's Hospital of Tampa, Tampa, Florida
  - Children's Memorial Hospital, Chicago, Illinois
  - Children's Hospital Boston, Boston, Massachusetts
  - Hackensack University Medical Center, Hackensack, New Jersey
  - St. Joseph's Children's Hospital, Paterson, New Jersey
  - The Brooklyn Hospital Center, Brooklyn, New York
  - Schneider Children's Hospital, New York, New York
  - SUNY - Upstate Medical University, Syracuse, New York
  - East Carolina University, Greenville, North Carolina
  - Akron Children's Hospital, Akron, Ohio
  - Children's Medical Center, Dayton, Ohio
  - Oklahoma State University Health Sciences Center, Oklahoma City, Oklahoma
  - Penn State University / Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - St. Jude Children's Research Hospital Memphis, Memphis, Tennessee
  - Cook's Children's Medical Center, Fort Worth, Texas
  - Texas Children's Hospital, Houston, Texas
  - Children's Hospital of the King's Daughters, Norfolk, Virginia